CLINICAL TRIAL: NCT07359144
Title: The Effect of Pilates Exercises on Nonspecific Low Back Pain in Postnatal Women
Brief Title: Pilates Exercises on Nonspecific Low Back Pain in Postnatal Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Eman Mosbah Mohamed Elsheikh, B.Sc. in Physical Therapy, Misr University for Science and Technology (2018), Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KFSIRB200-686
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Pilates Exercises; Nonspecific; Low Back Pain; Postnatal Women
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (A) (Study group): (Experimental): Patients will do a comprehensive exercise consisting of a home exercise program (bridges, bridge with leg extension (bridge dog), back extensions, spine twist, and child's pose), a Pilates program, and oral paracetamol as needed for pain relief.
  Interventions: Other: Pilates program + Home exercise program
- Group (B) (Control group) (Active Comparator): Patients will perform a home-based exercise program consisting solely of postural correction exercises.
  Interventions: Other: Home exercise program

INTERVENTIONS:
Other: Pilates program + Home exercise program — Patients will do a comprehensive exercise consisting of a home exercise program (bridges, bridge with leg extension (bridge dog), back extensions, spine twist, and child's pose), a Pilates program, and oral paracetamol as needed for pain relief.
  Arms: Group (A) (Study group):
Other: Home exercise program — Patients will perform a home-based exercise program consisting solely of postural correction exercises.
  Arms: Group (B) (Control group)

SUMMARY:
This study aims to investigate the effects of Pilates for postnatal women with Non-specific low back pain (NSLBP).

DETAILED DESCRIPTION:
Low back pain (LBP) is of high prevalence among adults, which can be related to factors such as sedentary lifestyle, being overweight or work conditions.

Non-specific LBP (NSLBP) is defined as pain in the lower back region that cannot be attributed to a recognizable, specific pathology such as infection, fracture, or nerve root compression.

Pilates exercises focus on improving core stability, flexibility, posture, and body awareness through controlled, precise movements. The integration of breathing techniques and concentration enhances the mind-body connection, which can contribute to pain reduction and functional improvement. For individuals with LBP, Pilates has been shown to improve strength and flexibility, reduce pain intensity, and enhance overall physical function, making it a promising intervention for managing musculoskeletal disorders.

ELIGIBILITY:
Inclusion Criteria:

* Age ranges from 20 and 30 years old.
* Body mass index (BMI) doesn't exceed 30 kg/m2.
* Patients who are referred from a gynecologist with a diagnosis of nonspecific low back pain.
* Patients who have pain for more than three months.
* Patients who have parity ranging from one to three (to control the extreme physiological changes from multiple childbirths, ensuring a more uniform sample).
* Patients who have score more than 4 on the Visual Analog Scale (VAS).

Exclusion Criteria:

* Mechanical low back pain (LBP).
* Women who had performed any spinal surgery e.g. unilateral hemilaminectomy or microdiscectomy.
* Women with history of vertebral fracture or trauma.
* Women with systemic disorder e.g. diabetes mellitus.
* Women who are pregnant.
* Women who had received physiotherapy treatment for their LBP one month before the start of this study.

Ages: 20 Years to 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Postnatal Women
Enrollment: 48 (Estimated)
Dates: Start 2026-01-22 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Pain Intensity | 3 months post-procedure
  Pain Intensity will be assessed using Visual Analog Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable").

SECONDARY OUTCOMES:
Assessment of pain pressure threshold | 3 months post-procedure
  Pain pressure threshold (PPT) will be determined using a handheld electronic pressure algometer with a 1 cm2 probe area with an increasing of the pressure rate of 20 Kpa/s. The pressure algometer consists of a "pistol" handle and a rod with a pressure-sensitive gauge strain at the tip.
Assessment of functional disability | 3 months post-procedure
  Oswestry Disability Index will be used to assess functional disability. It is a self-assessing questionnaire for low back pain, which includes 10 items; each contains six levels of answers ranging from 0-5. Its items include pain intensity, personal care, lifting objects, walking, sitting, standing, sleeping, sex life, social life, and travelling. A total score is calculated, divided by 50, and multiplied by 100. It ranges from 0% indicating no disability to 100% indicating complete disability.
Assessment of the quality of life | 3 months post-procedure
  Quality of life (QOL) will be assessed using SF-36 Questionnaire. SF-36 questionnaire consists of thirty-six questions measuring PH components (physical function, role physic, bodily pain, general health and MH components (vitality, social functioning, role emotion, general mental health). The response for each item was scored from 0-100, and the mean score of each domain was calculated. Lower score implied poor QoL, whereas higher score indicated excellent QoL.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University (Faculty of Physical Therapy), Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.